CLINICAL TRIAL: NCT01975090
Title: A Prospective, Multi-Center Study of the Novate Sentry Bioconvertible Vena Cava Filter
Brief Title: The SENTRY Clinical Study
Acronym: SENTRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Novate Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CI 036
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Results first posted 2017-10-12 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (1):
- SENTRY IVC Filter (Experimental): The SENTRY IVC Bioconvertible Filter
  Interventions: Device: SENTRY IVC Filter

INTERVENTIONS:
Device: SENTRY IVC Filter — The SENTRY IVC Bioconvertible Filter is designed to provide temporary protection to subjects at transient, high risk of pulmonary embolism. Following conclusion of the protection period The SENTRY filter bioconverts, and filter arms withdraw towards the IVC wall for incorporation; obviating the need for retrieval.

SUMMARY:
The SENTRY Bioconvertible Inferior Vena Cava (IVC) Filter has been developed to provide temporary protection against pulmonary embolism (PE).

DETAILED DESCRIPTION:
Pulmonary embolism (PE) is a prevalent disease with a significant morbidity and mortality. The estimated annual incidence is 1.45 per 1,000 patients, which translates to 1,350,000 cases per year in the United States. It is estimated that PE results in more than 200,000 deaths per year.

Currently there are two types of commercially available IVC filters utilized to prevent PE; permanent and retrievable. Both types of filters have documented limitations, such as tilting, migration, fracture, embolization and late deep vein thrombosis (DVT). Retrievable filters were developed to avert some of the late consequences of permanent filter, but in practice there is low success with eventual removal. In a series of 37 clinical studies, with a total of 6,834 patients the mean retrieval rate was 34%.

There are numerous design features of the SENTRY IVC Filter that are intended to improve on the limitations of available IVC filters and obviate the need for retrieval.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age
2. fully informed subject who has executed an Institutional Review Board (IRB) or Ethics Committee (EC) approved informed consent
3. willing and able to comply with follow-up visit requirements
4. requirement of transient PE protection of < 60 days
5. documented or high risk of PE or DVT
6. inability to use anti-coagulation due to contraindication, failure, complication or risk of injury from pharmacotherapy
7. IVC diameter compatible with filter diameter
8. IVC length adequate for filter placement

Exclusion Criteria:

1. intellectual impairment preventing understanding involvement in a clinical study
2. hypersensitivity to device components
3. impaired renal function defined as a serum creatinine level of > 2.0 mg/dL
4. active systemic infection
5. life expectancy < 12 months
6. malignancy extending PE risk > 60 days
7. pregnant or plans to become pregnant during study follow-up period
8. participating in another investigational trial that has not reached its primary endpoint
9. known hypercoaguable state
10. inherited or acquired hemostatic disorder
11. history or presence of a caval stent or filter
12. inability to gain femoral or jugular access
13. duplicated or left sided IVC
14. renal vein thrombosis or IVC thrombosis extending to the renal veins
15. jugular and femoral vein irregularity, stenosis or aneurysm that would interfere with successful device delivery
16. spinal irregularity that may interfere with successful device delivery
17. occlusive or free-floating thrombus in the IVC
18. contrast allergy that cannot be adequately pre-medicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Dake, MD, Principal Investigator — Stanford University
Locations (23):
- United States (20):
  - Brookwood Medical Center, Birmingham, Alabama
  - University of Alabama, Birmingham, Alabama
  - Stanford Hospital & Clinic, Palo Alto, California
  - Memorial Health System, Colorado Springs, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Adventist Midwest Health, Hinsdale, Illinois
  - St. Francis Hospital, Peoria, Illinois
  - Indiana University, Indianapolis, Indiana
  - Lakeview Regional Heart Center, Covington, Louisiana
  - Washington University in St Louis, St Louis, Missouri
  - Rutgers-New Jersey Medical School, Newark, New Jersey
  - University of North Carolina, Chapel Hill, North Carolina
  - Rex Hospital, Raleigh, North Carolina
  - Riverside Methodist Hospital, Columbus, Ohio
  - Jobst Vascular Institute, Toledo, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Texas Southwestern, Dallas, Texas
  - Providence Medical Research Center, Spokane, Washington
- Belgium (2):
  - Imelda Hospital, Bonheiden
  - AZ Sint-Blasius, Dendermonde
- Pontificia Universidad Catolica De Chile, Santiago, Chile

REFERENCES:
- [Background] Tsai AW, Cushman M, Rosamond WD, Heckbert SR, Polak JF, Folsom AR. Cardiovascular risk factors and venous thromboembolism incidence: the longitudinal investigation of thromboembolism etiology. Arch Intern Med. 2002 May 27;162(10):1182-9. doi: 10.1001/archinte.162.10.1182. PMID 12020191
- [Background] Grassi CJ, Swan TL, Cardella JF, Meranze SG, Oglevie SB, Omary RA, Roberts AC, Sacks D, Silverstein MI, Towbin RB, Lewis CA; Society of Cardiovascular & Interventional Radiology, Standards of Practice Committee. Quality improvement guidelines for percutaneous permanent inferior vena cava filter placement for the prevention of pulmonary embolism. SCVIR Standards of Practice Committee. J Vasc Interv Radiol. 2001 Feb;12(2):137-41. doi: 10.1016/s1051-0443(07)61818-1. No abstract available. PMID 11265876
- [Background] Angel LF, Tapson V, Galgon RE, Restrepo MI, Kaufman J. Systematic review of the use of retrievable inferior vena cava filters. J Vasc Interv Radiol. 2011 Nov;22(11):1522-1530.e3. doi: 10.1016/j.jvir.2011.08.024. PMID 22024114
- [Background] Morales JP, Li X, Irony TZ, Ibrahim NG, Moynahan M, Cavanaugh KJ Jr. Decision analysis of retrievable inferior vena cava filters in patients without pulmonary embolism. J Vasc Surg Venous Lymphat Disord. 2013 Oct;1(4):376-84. doi: 10.1016/j.jvsv.2013.04.005. Epub 2013 Jul 4. PMID 26992759
- [Background] Dake MD, Murphy TP, Kramer AH, Darcy MD, Sewall LE, Curi MA, Johnson MS, Arena F, Swischuk JL, Ansel GM, Silver MJ, Saddekni S, Brower JS, Mendes R; SENTRY Trial Investigators. One-Year Analysis of the Prospective Multicenter SENTRY Clinical Trial: Safety and Effectiveness of the Novate Sentry Bioconvertible Inferior Vena Cava Filter. J Vasc Interv Radiol. 2018 Oct;29(10):1350-1361.e4. doi: 10.1016/j.jvir.2018.05.009. Epub 2018 Sep 1. PMID 30177423
- [Background] Gaines PA, Kolodgie FD, Crowley G, Horan S, MacDonagh M, McLucas E, Rosenthal D, Strong A, Sweet M, Panchal DK. Sentry Bioconvertible Inferior Vena Cava Filter: Study of Stages of Incorporation in an Experimental Ovine Model. Int J Vasc Med. 2018 Jul 19;2018:6981505. doi: 10.1155/2018/6981505. eCollection 2018. PMID 30112213

RESULTS

PARTICIPANT FLOW:
Groups:
- SENTRY IVC Filter: Patients were enrolled with documented deep vein thrombosis (DVT) or PE or at temporary risk of developing DVT or PE, and unable to use anticoagulation.
Period: Overall Study
Arm/Group | SENTRY IVC Filter
Started | 129
6-month Follow-up | 117
Completed | 117
Not Completed | 12

BASELINE CHARACTERISTICS:
Groups:
- SENTRY IVC Filter Group: Patients were enrolled with documented deep vein thrombosis (DVT) or PE or at temporary risk of developing DVT or PE, and unable to use anticoagulation
Arm/Group | SENTRY IVC Filter Group
Number analyzed (Participants) | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 70
  >=65 years | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 73
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 4
  United States | 115
  Chile | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Reported Clinical Success
Description: A Composite Endpoint including:
  Technical success in deployment without acute Events; Freedom from Symptomatic Pulmonary Embolism; and Freedom from IVC filter related complications
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | SENTRY IVC Filter
Number analyzed (Participants) | 114
Participants | 111

2. Secondary Outcome: Number of Participants With IVC Filter Related Complications
Description: IVC filter related complications include, filter tilting, migration, embolization, fracture, vessel perforation, and symptomatic complications (symptomatic caval thrombosis, invasive filter intervention and filter-related death).
Time Frame: 6months
Population: Freedom from IVC Filter Related Complications was assessed by the site and reviewed by an Independent Core Lab. All subjects that had data collected were included in the analysis for population.
Measure: Number; unit: participants
Groups:
- Filter Tilting; Filter Migration; Filter Embolization; Filter Fracture; Filter Perforation: Core Lab reviewed imaging data at 6 month follow-up
- Symptomatic Complications: Symptomatic Complications is the composite of Symptomatic Caval Thrombosis and Other Symptomatic Complications Requiring Invasive Intervention and filter-related death at 6 months
Arm/Group | Filter Tilting | Filter Migration | Filter Embolization | Filter Fracture | Filter Perforation | Symptomatic Complications
Number analyzed (Participants) | 114 | 114 | 114 | 114 | 114 | 126
participants | 0 | 0 | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: 6 month adverse events were monitored by Organ Class .
Arm/Group | SENTRY IVC Filter
Serious Adverse Events (participants affected / at risk) | 45/129
Other Adverse Events (participants affected / at risk) | 85/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SENTRY IVC Filter (N=129)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 5
Cardiac disorders (Cardiac disorders) | 9
Gastrointestinal disorders (Gastrointestinal disorders) | 5
General disorders and administration site conditions (General disorders) | 3
Infections and infestations (Immune system disorders) | 18
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 4
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2
Neoplasms benign, malignant, and unspecified (including cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Nervous system disorders (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Psychiatric disorders (Psychiatric disorders) | 0
Renal and urinary disorders (Renal and urinary disorders) | 5
Respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 9
Vascular disorders (Vascular disorders) | 3
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0
Surgical and medical procedures (Surgical and medical procedures) | 0
Congenital, familial, and genetic disorders (Congenital, familial and genetic disorders) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SENTRY IVC Filter (N=129)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 13
Cardiac disorders (Cardiac disorders) | 19
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 19
General disorders and administration site conditions (General disorders) | 14
Infections and infestations (Infections and infestations) | 45
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 8
Investigations (Investigations) | 8
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 22
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 12
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Nervous system disorders (Nervous system disorders) | 17
Psychiatric disorders (Psychiatric disorders) | 7
Renal and urinary disorders (Renal and urinary disorders) | 16
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 26
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 5
Surgical and medical procedures (Surgical and medical procedures) | 6
Vascular disorders (Vascular disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No